CLINICAL TRIAL: NCT00312871
Title: Effect of Early Correction of Anemia on the Progression of Chronic Renal Insufficiency (ECAP)
Brief Title: Effects of Early Correction of Anemia in Patients With Chronic Renal Insufficiency
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped due to restrictions in labeling for the subcutaneous route of administration of EPREX.
Sponsor: Janssen Cilag S.A.S. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003181
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Renal Failure, Chronic Renal Failure
Keywords: Chronic renal failure; Anemia; Renal replacement therapy; Epoetin; Epoetin alfa; erythropoietin; Chronic kidney failure; end-stage renal disease
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of the study is to assess the effect of an early and complete correction of anemia after treatment with epoetin alfa on the rate of progression of chronic renal failure (which involves improper functioning of the kidneys). It also assesses the effect of hemoglobin normalization (correction of anemia) on the need for renal (kidney) replacement therapy, quality of life, blood pressure control, hospital admissions, mortality, cardiovascular events, nutritional status and safety.

DETAILED DESCRIPTION:
Epoetin alfa can increase hemoglobin levels in chronic renal failure patients (patients with persistent kidney dysfunction) resulting in minimal transfusion requirements and improved kidney function capacity. This study is a randomized (patients randomly divided into groups), multicenter, open-label (study drug is known to the patients) clinical trial to assess the effect of normalization of hemoglobin (defined as a hemoglobin level of 13-14 g/dL in women and 14-15 g/dL in men) on the rate of progression of chronic renal failure (persistent kidney dysfunction). The study duration is 40 months. The study is in two phases (Phase A = stabilization, Phase B = maintenance) with two patient groups (Group 1, Group 2) per phase. In Phase A (lasting 4 months) for patients in Group 1, hemoglobin is progressively increased to a target level. Phase A can be extended up to 6 months for Group 1 patients in whom the target hemoglobin (13-14 g/dL in women, 14-15 g/dL in men) is not reached. Patients in Group 2, hemoglobin is progressively increased up to 12 g/dL with epoetin alfa if it drops below 11 g/dL. For all patients in Phase A, Iron and vitamin deficiencies will also be corrected, and factors known to affect progression of renal failure (kidney dysfunction) will be optimized. In Phase B (lasting 36 months), effectiveness of anemia correction by epoetin alfa will be compared against non-correction (continued anemia) with regard to changes in kidney function. During this phase, patients will be maintained at the higher (Group 1) or lower (Group 2) target hemoglobin level. Safety data (including cardiovascular events, seizures, and hypertension) will be collected and monitored throughout the study. The hypothesis of the study is that correction of anemia may slow down kidney deterioration and progression of kidney failure to end-stage kidney disease that is caused by anemia-induced hypoxia, a state of oxygen deficiency in the kidney. Another hypothesis of the study is that genetic mutations (changes in the genes) may play a role in the progression of chronic renal failure. For those patients wishing to participate in this aspect of the study, blood samples will be collected for genomic DNA analysis and the results will be compiled to determine which genes are generally associated in the study population with kidney deterioration. Patients will receive epoetin alfa injections (25 to 100 IU/kg) under the skin 1 time per week. Dosage may be increased by 25 IU/kg increments to reach or maintain target hemoglobin, then dose maintained for study duration, as long as hemoglobin stays within range.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic renal failure, and at least a 6-month follow-up with at least 3 measurements of serum creatinine
* patients with a rate of decline in glomerular filtration rate (GFR--a measure of kidney function) below 0.6 mL/min/month
* patients with a hemoglobin level <13 g/dL for men and <12.5 g/dL for women without active blood loss or iron deficiency
* patients with a glomerular filtration rate (a measure of kidney function) between 25 and 60 mL/min/1.73m2)
* patients with blood pressure <=160/100 mm Hg (with or without antihypertensive therapy)

Exclusion Criteria:

* Patients with chronic renal failure (kidney dysfunction) associated with inherited polycystic kidney disease
* patients currently receiving treatment with epoetin for anemia secondary to chronic renal failure, and having a hemoglobin level >11 g/dL
* patients receiving epoetin but having a hemoglobin level below 11 g/dL will not be excluded
* patients with severe hypertension (blood pressure >= 180/110 mm Hg) within 3 months prior to study entry
* patients with a history of New York Heart Association (NYHA) class III or IV congestive heart failure within the preceding two years - NYHA class I and II congestive heart failure is accepted
* patients with a history of ischemic heart disease (deficient blood supply to the heart due to constricted or obstructed arteries)
* concurrent malignancy
* patients who have had a transfusion of red blood cells within 30 days prior to study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2001-02; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Rate of progression of chronic renal failure over 36 months as measured by at least 2 glomerular filtration rate assessments.

SECONDARY OUTCOMES:
Need for renal replacement therapy; quality of life; blood pressure control; hospital admissions; mortality; cardiovascular events; nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A.S. Clinical Trial, Study Director — Janssen Cilag S.A.S.

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: Effect of Early Correction Of Anaemia on the Progression of Chronic Renal Insufficiency (ECAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=273&filename=CR003181_CSR.pdf